CLINICAL TRIAL: NCT01455194
Title: Control of Moderate or Severe Asthma With 160, 320 and 640 mcg Ciclesonide/Day. A One-year Randomised, Double-blind, Multicenter Trial.
Brief Title: Effect of High Dose Ciclesonide on Asthma Control
Acronym: CONTRAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL-9709-301-RD; 2011-000683-99 (EudraCT Number); U1111-1133-6333 (Registry Identifier: WHO); CL-9709-301-RDCTID (Registry Identifier: Israel)
Record Dates: First submitted 2011-10-17; First posted 2011-10-19 (Estimated); Results first posted 2016-10-25 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Bronchial Asthma
Keywords: ciclesonide; asthma
MeSH Terms: conditions — Asthma | interventions — ciclesonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- CIC 160 (Active Comparator): Two puffs of 40 mcg ciclesonide inhaled in the morning and the evening (corresponding to a total daily dose of 160 mcg)
  Interventions: Drug: Ciclesonide
- CIC 320 (Active Comparator): Two puffs of 80 mcg ciclesonide inhaled in the morning and the evening (corresponding to a total daily dose of 320 mcg)
  Interventions: Drug: Ciclesonide
- CIC 640 (Active Comparator): Two puffs of 160 mcg ciclesonide inhaled in the morning and the evening (corresponding to a total daily dose of 640 mcg)
  Interventions: Drug: Ciclesonide

INTERVENTIONS:
Drug: Ciclesonide — During the treatment period subjects will inhale two puffs of either 40, 80 or 160 μg ciclesonide in the morning and the evening (corresponding to a total daily dose of 160, 320 or 640 μg)

SUMMARY:
The aim of the trial is to investigate asthma control with 160 to 640 mcg ciclesonide/day. Asthma control will be assessed by the Asthma Control Questionnaire (ACQ).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent was provided
* History of persistent bronchial asthma for at least 6 months
* Current treatment with an Inhaled Corticosteroid (ICS) at a stable dose in the dose range of 200-1000 μg Fluticasone Propionate (FP)/day or equivalent for a minimum of 12 weeks
* Good inhalation technique
* Under the current ICS pre-treatment the ACQ score ranges between ≥ 0.75 and ≥ 2

Exclusion Criteria:

* Clinically relevant abnormal laboratory values suggesting an unknown disease and requiring further clinical evaluation
* Concomitant severe diseases (e.g. malignant diseases during the past 5 years [other than basal or squamous cell carcinoma], hepatitis C, acquired immune deficiency syndrome [AIDS])
* Diseases which are contraindications for the use of ICS (e.g. active or inactive pulmonary tuberculosis or relevant fungal, bacterial or viral infections of the lower respiratory tract demanding specific treatment)
* Use of systemic glucocorticosteroids within 4 weeks (injectable depot steroids 6 weeks) before entry into the baseline period, or more than 3 times during the last 6 months

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2011-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (30):
- Argentina (6):
  - Buenos Aires
  - Capital Federal, Buenos Aires
  - Rosario
  - Rosario-Santa Fe
  - Salta
  - San Miguel de Tucumán
- Brazil (7):
  - Florianópolis
  - Goiânia
  - Porto Alegre
  - Rio de Janiero
  - Santo André
  - São Paulo
  - Sorocaba
- Germany (5):
  - Berlin
  - Bonn
  - Landsberg
  - Rüdersdorf
  - Schwetzingen
- Israel (7):
  - Beersheba
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Rehovot
  - Tel Aviv
- Russia (5):
  - Barnaul
  - Moscow
  - Novosibirsk
  - Saint Petersburg
  - Tomsk

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in Argentina, Brazil, Germany, Israel and Russia from 10 November 2011 to 15 August 2014.
Pre-assignment Details: Participants with a historical diagnosis of persistent bronchial asthma for at least 6 months,treated with a stable inhaled corticosteroid (ICS)dose for at least 12 weeks were enrolled in a single-blind baseline period receiving 160 microgram(mcg)ciclesonide,then a double-blind treatment period in 1 of 3 treatment arms: ciclesonide 160,320,640 mcg.
Groups:
- Baseline Period: Ciclesonide 160 mcg: Ciclesonide 80 mcg, metered dose inhaler (MDI), inhalational, twice daily for up to 3 weeks in the baseline period.
- Treatment Period: Ciclesonide 160 mcg: Ciclesonide 80 mcg, metered dose inhaler (MDI), inhalational, twice daily for up to 3 weeks in the baseline period. Ciclesonide 80 mcg, MDI, inhalational, twice daily for up to 52 weeks in the double blind treatment period.
- Treatment Period: Ciclesonide 320 mcg: Ciclesonide 160 mcg, MDI, inhalational, twice daily for up to 52 weeks in the double blind treatment period.
- Treatment Period: Ciclesonide 640 mcg: Ciclesonide 320 mcg, MDI, inhalational, twice daily for up to 52 weeks in the double blind treatment period.
Period: Overall Study
Arm/Group | Baseline Period: Ciclesonide 160 mcg | Treatment Period: Ciclesonide 160 mcg | Treatment Period: Ciclesonide 320 mcg | Treatment Period: Ciclesonide 640 mcg
Started | 153 | 120 | 122 | 125
Completed | 0 | 89 | 92 | 97
Not Completed | 153 | 31 | 30 | 28
Not completed — Screen Failure | 20 | 0 | 0 | 0
Not completed — Randomisation Failure | 90 | 0 | 0 | 0
Not completed — Deterioration in asthma | 12 | 6 | 14 | 9
Not completed — Adverse Event | 1 | 1 | 1 | 3
Not completed — Withdrawal by Subject | 21 | 16 | 12 | 9
Not completed — Lost to Follow-up | 2 | 0 | 1 | 1
Not completed — Pregnancy | 0 | 1 | 1 | 0
Not completed — Discontinuation criterion fulfilled | 3 | 2 | 0 | 2
Not completed — Miscellaneous | 4 | 5 | 1 | 4

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) was defined as all randomized participants who took at least 1 dose of double-blind study medication.Baseline data was summarized only for those participants who entered treatment period which was the core period of the trial.
Groups:
- Treatment Period: Ciclesonide 160 mcg: Ciclesonide 80 mcg, MDI, inhalational, twice daily for up to 52 weeks in the double blind treatment period.
- Total: Total of all reporting groups
Arm/Group | Treatment Period: Ciclesonide 160 mcg | Treatment Period: Ciclesonide 320 mcg | Treatment Period: Ciclesonide 640 mcg | Total
Number analyzed (Participants) | 120 | 122 | 125 | 367
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (14.86) | 44.7 (15.60) | 45.3 (16.22) | 44.4 (15.57)
Gender [Count of Participants; unit: Participants]
  Female | 72 | 77 | 81 | 230
  Male | 48 | 45 | 44 | 137
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 6 | 5 | 4 | 15
  White | 113 | 115 | 114 | 342
  Unknown or Not Reported | 1 | 2 | 7 | 10
Height [Mean (Standard Deviation); unit: meter (m)] | 1.65 (0.093) | 1.66 (0.101) | 1.65 (0.104) | 1.65 (0.099)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 74.59 (16.371) | 77.98 (18.993) | 73.72 (14.660) | 75.42 (16.811)
Body Mass Index [Mean (Standard Deviation); unit: kilogram per meter square (kg/m^2)] | 27.34 (5.217) | 28.42 (6.346) | 27.12 (5.373) | 27.62 (5.681)
History of exacerbations [Number; unit: participants] — Asthma exacerbations were defined as a worsening of asthma requiring either treatment with oral (or other systemic) glucocorticosteroids for at least 3 days or hospitalisation or a visit to the emergency room because of asthma.
  participants
    0 | 70 | 70 | 63 | 203
    1 | 17 | 19 | 21 | 57
    2-3 | 4 | 3 | 4 | 11
    4+ | 0 | 0 | 0 | 0
    Unknown | 29 | 30 | 37 | 96
Smoking Status [Number; unit: participants]
  Never | 109 | 102 | 109 | 320
  Current | 1 | 1 | 1 | 3
  Former | 10 | 19 | 15 | 44
Prestudy ICS dose [Number; unit: participants]
  <200(mcg/day) fluticasone propionate(FP)equivalent | 3 | 3 | 2 | 8
  Low:>=200 mcg/day(=<)250 mcg/day FP equivalent | 40 | 37 | 42 | 119
  Medium:>250 mcg/dayto=<500 mcg/day FP equivalent | 72 | 75 | 70 | 217
  High:>500 mcg/dayto=<1000 mcg/day FP equivalent | 5 | 7 | 11 | 23
Baseline asthma control questionnaire (ACQ) [Mean (Standard Deviation); unit: units on scale] — ACQ=5 questions about symptoms,1 question about beta 2-agonist use and 1 about lung function (FEV1% predicted).Participants recall their experiences during the previous 7 days and respond to each question using a 7-point scale.The items are equally weighted and the ACQ score is the mean of 7 items and ranges between 0 (well controlled) and 6 (extremely poorly controlled). Mean scores of =<0.75 indicate well-controlled asthma, scores between 0.76 and < 1.5 indicate partly controlled asthma, and a score >= 1.5 indicates uncontrolled asthma.
  units on scale | 2.24 (0.304) | 2.16 (0.384) | 2.20 (0.361) | 2.20 (0.363)
Pre-forced expiratory volume in 1 second (FEV1) [Mean (Standard Deviation); unit: liter (L)] — Pre-FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration prior to salbutamol administration.
  liter (L) | 2.20 (0.792) | 2.35 (0.798) | 2.23 (0.801) | 2.26 (0.797)
Post-FEV1 [Mean (Standard Deviation); unit: L] — Post-FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration after salbutamol administration.
  L | 2.71 (0.915) | 2.84 (0.883) | 2.76 (0.906) | 2.77 (0.900)
FEV1 reversibility [Mean (Standard Deviation); unit: percent reversibility] — Reversibility is assessed using FEV1 measurements. Percent reversibility is calculated as the difference between highest FEV1 after salbutamol and highest FEV 1 before salbutamol divided by highest FEV 1 before salbutamol. FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration.
  percent reversibility | 25.5 (17.02) | 23 (17.10) | 26.5 (20.78) | 25.0 (18.41)
Pre FEV1 predicted [Mean (Standard Deviation); unit: percent of predicted] — Pre-FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration prior to salbutamol administration. It is converted to the percentage of predicted FEV1 based on age, gender, weight and race of participants. Generally, values between 80% to 120% are considered normal.
  percent of predicted | 69.095 (18.4683) | 74.345 (16.7285) | 71.835 (18.4365) | 71.773 (17.9737)
Post FEV1 predicted [Mean (Standard Deviation); unit: percent of predicted] — Post-FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration after salbutamol administration. It is converted to the percentage of predicted FEV1 based on age, gender, weight and race of participants. Generally, values between 80% to 120% are considered normal.
  percent of predicted | 84.893 (19.3038) | 90.168 (17.7365) | 88.505 (17.7105) | 87.875 (18.3373)

OUTCOME MEASURES:

1. Primary Outcome: Asthma Control Questionnaire (ACQ) Score at Baseline
Description: The ACQ was developed to measure the adequacy of asthma control in clinical research and in clinical practice. It includes 5 questions about symptoms, 1 question about beta 2 -agonist use and 1 about lung function (FEV1% predicted). Participants recall their experiences during the previous 7 days and respond to each question using a 7-point scale. The items are equally weighted and the ACQ score is the mean of 7 items and ranges between 0 (well controlled) and 6 (extremely poorly controlled). Mean scores of =<0.75 indicate well-controlled asthma, scores between 0.76 and < 1.5 indicate partly controlled asthma, and a score >= 1.5 indicates uncontrolled asthma.
Time Frame: Baseline
Population: The intent-to-treat (ITT) analysis set included participants having at least 1 postrandomization efficacy assessment.This outcome measure was planned to be analyzed on for the treatment period.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Treatment Period: Ciclesonide 160 mcg | Treatment Period: Ciclesonide 320 mcg | Treatment Period: Ciclesonide 640 mcg
Number analyzed (Participants) | 120 | 119 | 122
units on a scale | 2.24 (0.031) | 2.15 (0.035) | 2.19 (0.032)

2. Primary Outcome: Change From Baseline in ACQ Score to Tlast
Description: as for outcome 1
Time Frame: Week 52
Population: The ITT analysis set included participants having at least 1 postrandomization efficacy assessment.This outcome measure was planned to be analyzed on for the treatment period.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Treatment Period: Ciclesonide 160 mcg | Treatment Period: Ciclesonide 320 mcg | Treatment Period: Ciclesonide 640 mcg
Number analyzed (Participants) | 120 | 119 | 122
units on a scale | -0.833 (0.1028) | -0.799 (0.1019) | -0.955 (0.0969)
Statistical Analysis 1: Comparison: Treatment Period: Ciclesonide 160 mcg vs Treatment Period: Ciclesonide 640 mcg; Least square (LS) mean difference were derived from an ANCOVA model with baseline ACQ and age as covariates, and treatment, centre pool, sex, and prestudy ICS dose as factors; Test type: Superiority or Other; p = 0.2988, ANCOVA; LS Mean Difference = -0.122, 95% CI 2-sided [-0.353 to 0.109], Standard Error of Mean 0.1175
Statistical Analysis 2: Comparison: Treatment Period: Ciclesonide 160 mcg vs Treatment Period: Ciclesonide 320 mcg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.7741, ANCOVA; LS Mean Difference = 0.034, 95% CI 2-sided [-0.198 to 0.266], Standard Error of Mean 0.1180
Statistical Analysis 3: Comparison: Treatment Period: Ciclesonide 320 mcg vs Treatment Period: Ciclesonide 640 mcg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1835, ANCOVA; LS Mean Difference = -0.156, 95% CI 2-sided [-0.387 to 0.074], Standard Error of Mean 0.1172

3. Secondary Outcome: Time Course of ACQ
Description: The time course of the incidence of a 0.5 points improvement of ACQ score was evaluated. Mean ACQ values over time by treatment group for on-treatment site measurements was assessed. The time course of asthma control (ACQ) was done on a weekly base using home-based and site-based ACQ measurements. The ACQ was developed to measure the adequacy of asthma control in clinical research and in clinical practice. It includes 5 questions about symptoms, 1 question about beta 2 -agonist use and 1 about lung function (FEV1% predicted). Participants recall their experiences during the previous 7 days and respond to each question using a 7-point scale. The items are equally weighted and the ACQ score is the mean of 7 items and ranges between 0 (well controlled) and 6 (extremely poorly controlled). Mean scores of =<0.75 indicate well-controlled asthma, scores between 0.76 and < 1.5 indicate partly controlled asthma, and a score >= 1.5 indicates uncontrolled asthma.
Time Frame: Baseline, Week 52 (Treatment period)
Population: as for outcome 2
Measure: Median (Full Range); unit: Weeks
Arm/Group | Treatment Period: Ciclesonide 160 mcg | Treatment Period: Ciclesonide 320 mcg | Treatment Period: Ciclesonide 640 mcg
Number analyzed (Participants) | 105 | 108 | 115
Weeks | 1.100 [0.00 to 4.40] | 1.000 [0.00 to 3.90] | 1.000 [0.00 to 4.60]

4. Secondary Outcome: Number of Weeks With Well-controlled Asthma Over the Course of the Study
Description: The number of weeks with well-controlled asthma is defined as the number of weeks that the participant had an ACQ score of 0.75 or lower over the course of the study. The ACQ was developed to measure the adequacy of asthma control in clinical research and in clinical practice. It includes 5 questions about symptoms, 1 question about beta 2 -agonist use and 1 about lung function (FEV1% predicted). Participants recall their experiences during the previous 7 days and respond to each question using a 7-point scale. The items are equally weighted and the ACQ score is the mean of 7 items and ranges between 0 (well controlled) and 6 (extremely poorly controlled). Mean scores of =<0.75 indicate well-controlled asthma, scores between 0.76 and < 1.5 indicate partly controlled asthma, and a score >= 1.5 indicates uncontrolled asthma.
Time Frame: Baseline up to Week 52 (treatment period)
Population: The intent-to-treat ITT analysis set included participants having at least 1 postrandomization efficacy assessment.This outcome measure was planned to be analyzed on for the treatment period.
Measure: Number; unit: weeks
Units Other Than Participants: weeks
Arm/Group | Treatment Period: Ciclesonide 160 mcg | Treatment Period: Ciclesonide 320 mcg | Treatment Period: Ciclesonide 640 mcg
Number analyzed (Participants) | 120 | 119 | 122
Number analyzed (weeks) | 5286 | 5388 | 5669
weeks | 1211 | 1514 | 1447
Statistical Analysis 1: Comparison: Treatment Period: Ciclesonide 160 mcg vs Treatment Period: Ciclesonide 640 mcg; Test type: Superiority or Other; p = 0.8465, Wilcoxon (Mann-Whitney); Hodges-Lehmann point estimate = 0.000, 95% CI 2-sided [-3.000 to 4.000] — Treatment comparisons were carried out using an exact Wilcoxon Mann Whitney test
Statistical Analysis 2: Comparison: Treatment Period: Ciclesonide 160 mcg vs Treatment Period: Ciclesonide 320 mcg; Test type: Superiority or Other; p = 0.4175, Wilcoxon (Mann-Whitney); Hodges-Lehmann point estimate = 1.000, 95% CI 2-sided [-2.000 to 5.000] — Treatment comparisons were carried out using an exact Wilcoxon Mann Whitney test

5. Secondary Outcome: Number of Participants With Well-controlled Asthma and ACQ Improvement at the End of the Study
Description: Well-controlled asthma at the end of the study was defined as a participant with an ACQ score of 0.75 or lower. ACQ improvement was defined as a decrease in ACQ score of at least 0.5. The ACQ was developed to measure the adequacy of asthma control in clinical research and in clinical practice. It includes 5 questions about symptoms, 1 question about beta 2 -agonist use and 1 about lung function (FEV1% predicted). Participants recall their experiences during the previous 7 days and respond to each question using a 7-point scale. The items are equally weighted and the ACQ score is the mean of 7 items and ranges between 0 (well controlled) and 6 (extremely poorly controlled). Mean scores of =<0.75 indicate well-controlled asthma, scores between 0.76 and < 1.5 indicate partly controlled asthma, and a score >= 1.5 indicates uncontrolled asthma.
Time Frame: Week 52
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Treatment Period: Ciclesonide 160 mcg | Treatment Period: Ciclesonide 320 mcg | Treatment Period: Ciclesonide 640 mcg
Number analyzed (Participants) | 120 | 122 | 125
participants
  Well-controlled Asthma | 38 | 45 | 51
  ACQ Improvement | 87 | 81 | 85
Statistical Analysis 1: Comparison: Treatment Period: Ciclesonide 160 mcg vs Treatment Period: Ciclesonide 320 mcg; Well-controlled Asthma; Test type: Superiority or Other; p = 0.4186, Fisher Exact
Statistical Analysis 2: Comparison: Treatment Period: Ciclesonide 160 mcg vs Treatment Period: Ciclesonide 640 mcg; Well-controlled Asthma; Test type: Superiority or Other; p = 0.1460, Fisher Exact
Statistical Analysis 3: Comparison: Treatment Period: Ciclesonide 320 mcg vs Treatment Period: Ciclesonide 640 mcg; Well-controlled Asthma; Test type: Superiority or Other; p = 0.6017, Fisher Exact
Statistical Analysis 4: Comparison: Treatment Period: Ciclesonide 160 mcg vs Treatment Period: Ciclesonide 320 mcg; ACQ Improvement; Test type: Superiority or Other; p = 0.3305, Fisher Exact
Statistical Analysis 5: Comparison: Treatment Period: Ciclesonide 160 mcg vs Treatment Period: Ciclesonide 640 mcg; ACQ Improvement; Test type: Superiority or Other; p = 0.4860, Fisher Exact
Statistical Analysis 6: Comparison: Treatment Period: Ciclesonide 320 mcg vs Treatment Period: Ciclesonide 640 mcg; ACQ Improvement; Test type: Superiority or Other; p = 0.8922, Fisher Exact

6. Secondary Outcome: Number of Participants Reporting Time to First Well-Controlled Asthma and ACQ Improvement
Description: as for outcome 5
Time Frame: Baseline up to Week 52 (treatment period)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Treatment Period: Ciclesonide 160 mcg | Treatment Period: Ciclesonide 320 mcg | Treatment Period: Ciclesonide 640 mcg
Number analyzed (Participants) | 120 | 122 | 125
participants
  Well-controlled Asthma | 73 | 84 | 81
  ACQ Improvement | 112 | 107 | 115
Statistical Analysis 1: Comparison: Treatment Period: Ciclesonide 160 mcg vs Treatment Period: Ciclesonide 640 mcg; Well-controlled Asthma; Test type: Superiority or Other; p = 0.6062, Log Rank; Hazard Ratio (HR) = 1.042, 95% CI 2-sided [0.890 to 1.221], Standard Error of Mean 0.0806 — A hazard ratio of >1 represented a benefit for the test treatment
Statistical Analysis 2: Comparison: Treatment Period: Ciclesonide 160 mcg vs Treatment Period: Ciclesonide 640 mcg; ACQ Improvement; Test type: Superiority or Other; p = 0.4674, Log Rank; Hazard Ratio (HR) = 1.050, 95% CI 2-sided [0.921 to 1.197], Standard Error of Mean 0.0669 — A hazard ratio of >1 represented a benefit for the test treatment
Statistical Analysis 3: Comparison: Treatment Period: Ciclesonide 160 mcg vs Treatment Period: Ciclesonide 320 mcg; Well-controlled Asthma; Test type: Superiority or Other; p = 0.2523, Log Rank; Hazard Ratio (HR) = 1.201, 95% CI 2-sided [0.878 to 1.642], Standard Error of Mean 0.1597 — A hazard ratio of >1 represented a benefit for the test treatment
Statistical Analysis 4: Comparison: Treatment Period: Ciclesonide 160 mcg vs Treatment Period: Ciclesonide 320 mcg; ACQ Improvement; Test type: Superiority or Other; p = 0.5026, Log Rank; Hazard Ratio (HR) = 0.913, 95% CI 2-sided [0.700 to 1.191], Standard Error of Mean 0.1354 — A hazard ratio of >1 represented a benefit for the test treatment
Statistical Analysis 5: Comparison: Treatment Period: Ciclesonide 320 mcg vs Treatment Period: Ciclesonide 640 mcg; Well-controlled Asthma; Test type: Superiority or Other; p = 0.4893, Log Rank; Hazard Ratio (HR) = 0.898, 95% CI 2-sided [0.661 to 1.219], Standard Error of Mean 0.1560 — A hazard ratio of >1 represented a benefit for the test treatment
Statistical Analysis 6: Comparison: Treatment Period: Ciclesonide 320 mcg vs Treatment Period: Ciclesonide 640 mcg; ACQ Improvement; Test type: Superiority or Other; p = 0.2193, Log Rank; Hazard Ratio (HR) = 1.181, 95% CI 2-sided [0.906 to 1.538], Standard Error of Mean 0.1351 — A hazard ratio of >1 represented a benefit for the test treatment

7. Secondary Outcome: Number of Participants Reporting Time to First Well-Controlled Asthma Measurement by ACQ Cut-Off Point
Description: Well-controlled asthma was defined as an ACQ score of equal to or lower than the ACQ cut-off point.The ACQ was developed to measure the adequacy of asthma control in clinical research and in clinical practice. It includes 5 questions about symptoms, 1 question about beta 2 -agonist use and 1 about lung function (FEV1% predicted). Participants recall their experiences during the previous 7 days and respond to each question using a 7-point scale. The items are equally weighted and the ACQ score is the mean of 7 items and ranges between 0 (well controlled) and 6 (extremely poorly controlled). Mean scores of =<0.75 indicate well-controlled asthma, scores between 0.76 and < 1.5 indicate partly controlled asthma, and a score >= 1.5 indicates uncontrolled asthma.
Time Frame: Baseline up to Week 52 (treatment period)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Treatment Period: Ciclesonide 160 mcg | Treatment Period: Ciclesonide 320 mcg | Treatment Period: Ciclesonide 640 mcg
Number analyzed (Participants) | 120 | 122 | 125
participants
  ACQ cut-off at 0.5 | 56 | 69 | 63
  ACQ cut-off at 1.0 | 91 | 95 | 93
  ACQ cut-off at 1.25 | 99 | 101 | 101
  ACQ cut-off at 1.5 | 103 | 105 | 107
Statistical Analysis 1: Comparison: Treatment Period: Ciclesonide 160 mcg vs Treatment Period: Ciclesonide 640 mcg; ACQ cut-off at 0.5; Test type: Superiority or Other; p = 0.5397, Log Rank; Hazard Ratio (HR) = 1.058, 95% CI 2-sided [0.884 to 1.266], Standard Error of Mean 0.0917 — A hazard ratio of >1 represented a benefit for the test treatment
Statistical Analysis 2: Comparison: Treatment Period: Ciclesonide 160 mcg vs Treatment Period: Ciclesonide 640 mcg; ACQ cut-off at 1.0; Test type: Superiority or Other; p = 0.9458, Log Rank; Hazard Ratio (HR) = 1.005, 95% CI 2-sided [0.870 to 1.161], Standard Error of Mean 0.0738 — A hazard ratio of >1 represented a benefit for the test treatment
Statistical Analysis 3: Comparison: Treatment Period: Ciclesonide 160 mcg vs Treatment Period: Ciclesonide 640 mcg; ACQ cut-off at 1.25; Test type: Superiority or Other; p = 0.7213, Log Rank; Hazard Ratio (HR) = 1.026, 95% CI 2-sided [0.893 to 1.178], Standard Error of Mean 0.0708 — A hazard ratio of >1 represented a benefit for the test treatment
Statistical Analysis 4: Comparison: Treatment Period: Ciclesonide 160 mcg vs Treatment Period: Ciclesonide 640 mcg; ACQ cut-off at 1.5; Test type: Superiority or Other; p = 0.4807, Log Rank; Hazard Ratio (HR) = 1.050, 95% CI 2-sided [0.917 to 1.202], Standard Error of Mean 0.0692 — A hazard ratio of >1 represented a benefit for the test treatment
Statistical Analysis 5: Comparison: Treatment Period: Ciclesonide 160 mcg vs Treatment Period: Ciclesonide 320 mcg; ACQ cut-off at 0.5; Test type: Superiority or Other; p = 0.1150, Log Rank; Hazard Ratio (HR) = 1.326, 95% CI 2-sided [0.934 to 1.884], Standard Error of Mean 0.1791 — A hazard ratio of >1 represented a benefit for the test treatment
Statistical Analysis 6: Comparison: Treatment Period: Ciclesonide 160 mcg vs Treatment Period: Ciclesonide 320 mcg; ACQ cut-off at 1.0; Test type: Superiority or Other; p = 0.6281, Log Rank; Hazard Ratio (HR) = 1.074, 95% CI 2-sided [0.805 to 1.431], Standard Error of Mean 0.1467 — A hazard ratio of >1 represented a benefit for the test treatment
Statistical Analysis 7: Comparison: Treatment Period: Ciclesonide 160 mcg vs Treatment Period: Ciclesonide 320 mcg; ACQ cut-off at 1.25; Test type: Superiority or Other; p = 0.6853, Log Rank; Hazard Ratio (HR) = 1.059, 95% CI 2-sided [0.803 to 1.397], Standard Error of Mean 0.1415 — A hazard ratio of >1 represented a benefit for the test treatment
Statistical Analysis 8: Comparison: Treatment Period: Ciclesonide 160 mcg vs Treatment Period: Ciclesonide 320 mcg; ACQ cut-off at 1.5; Test type: Superiority or Other; p = 0.6995, Log Rank; Hazard Ratio (HR) = 1.055, 95% CI 2-sided [0.804 to 1.385], Standard Error of Mean 0.1388 — A hazard ratio of >1 represented a benefit for the test treatment
Statistical Analysis 9: Comparison: Treatment Period: Ciclesonide 320 mcg vs Treatment Period: Ciclesonide 640 mcg; ACQ cut-off at 0.5; Test type: Superiority or Other; p = 0.3080, Log Rank; Hazard Ratio (HR) = 0.837, 95% CI 2-sided [0.595 to 1.178], Standard Error of Mean 0.1744 — A hazard ratio of >1 represented a benefit for the test treatment
Statistical Analysis 10: Comparison: Treatment Period: Ciclesonide 320 mcg vs Treatment Period: Ciclesonide 640 mcg; ACQ cut-off at 1.0; Test type: Superiority or Other; p = 0.6645, Log Rank; Hazard Ratio (HR) = 0.939, 95% CI 2-sided [0.705 to 1.250], Standard Error of Mean 0.1461 — A hazard ratio of >1 represented a benefit for the test treatment
Statistical Analysis 11: Comparison: Treatment Period: Ciclesonide 320 mcg vs Treatment Period: Ciclesonide 640 mcg; ACQ cut-off at 1.25; Test type: Superiority or Other; p = 0.9564, Log Rank; Hazard Ratio (HR) = 0.992, 95% CI 2-sided [0.753 to 1.308], Standard Error of Mean 0.1408 — A hazard ratio of >1 represented a benefit for the test treatment
Statistical Analysis 12: Comparison: Treatment Period: Ciclesonide 320 mcg vs Treatment Period: Ciclesonide 640 mcg; ACQ cut-off at 1.5; Test type: Superiority or Other; p = 0.7367, Log Rank; Hazard Ratio (HR) = 1.047, 95% CI 2-sided [0.800 to 1.371], Standard Error of Mean 0.1375 — A hazard ratio of >1 represented a benefit for the test treatment

8. Secondary Outcome: Number of Participants Reporting Time to First Asthma Exacerbation
Description: Asthma exacerbations were defined as a worsening of asthma requiring either treatment with oral (or other systemic) glucocorticosteroids for at least 3 days or hospitalisation or a visit to the emergency room because of asthma. Baseline was defined as the average of the ACQ measurements of the last 2 weeks at site prior to first intake of double-blind study medication
Time Frame: Baseline up to Week 52 (treatment period)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Treatment Period: Ciclesonide 160 mcg | Treatment Period: Ciclesonide 320 mcg | Treatment Period: Ciclesonide 640 mcg
Number analyzed (Participants) | 120 | 122 | 125
participants | 5 | 11 | 10
Statistical Analysis 1: Comparison: Treatment Period: Ciclesonide 160 mcg vs Treatment Period: Ciclesonide 640 mcg; Test type: Superiority or Other; p = 0.2264, Log Rank; Hazard Ratio (HR) = 1.367, 95% CI 2-sided [0.824 to 2.267], Standard Error of Mean 0.2583 — A hazard ratio of <1 represented a benefit for the test treatment
Statistical Analysis 2: Comparison: Treatment Period: Ciclesonide 160 mcg vs Treatment Period: Ciclesonide 320 mcg; Test type: Superiority or Other; p = 0.1373, Log Rank; Hazard Ratio (HR) = 2.102, 95% CI 2-sided [0.789 to 5.602], Standard Error of Mean 0.5001 — A hazard ratio of <1 represented a benefit for the test treatment
Statistical Analysis 3: Comparison: Treatment Period: Ciclesonide 320 mcg vs Treatment Period: Ciclesonide 640 mcg; Test type: Superiority or Other; p = 0.7732, Log Rank; Hazard Ratio (HR) = 0.882, 95% CI 2-sided [0.375 to 2.074], Standard Error of Mean 0.4365 — A hazard ratio of <1 represented a benefit for the test treatment

9. Secondary Outcome: Number of Participants Reporting Asthma Exacerbations Rates
Description: Participants with at least 1 asthma exacerbation in the double-blind treatment period have been reported. As predefined in the protocol, the results for participants with missing data for any category were not included.
Time Frame: Baseline up to Week 52 (treatment period)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Treatment Period: Ciclesonide 160 mcg | Treatment Period: Ciclesonide 320 mcg | Treatment Period: Ciclesonide 640 mcg
Number analyzed (Participants) | 120 | 122 | 122
participants | 5 | 10 | 10
Statistical Analysis 1: Comparison: Treatment Period: Ciclesonide 160 mcg vs Treatment Period: Ciclesonide 640 mcg; Test type: Superiority or Other; p = 0.2880, Fisher Exact
Statistical Analysis 2: Comparison: Treatment Period: Ciclesonide 160 mcg vs Treatment Period: Ciclesonide 320 mcg; Test type: Superiority or Other; p = 0.2864, Fisher Exact

10. Secondary Outcome: Number of Participants With Markedly High Benefits
Description: The analyses was intended to identify participant's subsets that would benefit from dose escalation. This analysis tested the potential factors, including age, sex, pretrial inhaled corticosteroid (ICS) dose category, history of exacerbations, baseline ACQ score, baseline BMI category and smoking status. ACQ includes 5 questions about symptoms, 1 about beta 2 -agonist use and 1 about lung function (FEV1% predicted). Participants recall their experiences during the previous 7 days and respond to each question using a 7-point scale. The items are equally weighted and the ACQ score is the mean of 7 items and ranges between 0 (well controlled) and 6 (extremely poorly controlled).Mean scores of =<0.75 indicate well-controlled asthma, scores between 0.76 and < 1.5 indicate partly controlled asthma, and a score >=1.5 indicates uncontrolled asthma. As predefined in the protocol, participants with missing data for any category were not included.
Time Frame: Week 1 up to Week 52
Population: Safety analysis set included all participants who took at least 1 dose of study medication.One participant erroneously randomized into 160 mcg arm, actually received 640 mcg dose.For safety analysis, participants were analyzed based on the treatment they actually received.
Measure: Number; unit: participants
Arm/Group | Treatment Period: Ciclesonide 160 mcg | Treatment Period: Ciclesonide 320 mcg | Treatment Period: Ciclesonide 640 mcg
Number analyzed (Participants) | 119 | 122 | 126
participants | 0 | 0 | 0

11. Secondary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAE)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. TEAE is defined as an adverse event with an onset that occurs after receiving study drug. AEs included both serious AEs and non-serious AEs. Baseline of double-blind treatment period was defined as the average of the measurements of the last 2 weeks at site prior to first intake of double-blind study medication.
Time Frame: Baseline period (Week -3 up to -1), treatment period (Baseline up to Week 56)
Population: as for outcome 10
Measure: Number; unit: participants
Groups:
- Baseline Period: Ciclesonide 160 mcg: Ciclesonide 80 mcg, MDI, inhalational, twice daily for up to 3 weeks in the baseline period.
Arm/Group | Baseline Period: Ciclesonide 160 mcg | Treatment Period: Ciclesonide 160 mcg | Treatment Period: Ciclesonide 320 mcg | Treatment Period: Ciclesonide 640 mcg
Number analyzed (Participants) | 520 | 119 | 122 | 126
participants | 109 | 85 | 86 | 89

12. Secondary Outcome: Number of Participants Reporting Clinically Significant Change From Baseline in Vital Signs
Description: Vital signs included body temperature, blood pressure (BP) and pulse rate. Normal range for vital signs included: Systolic BP >170 millimeters of mercury (mm Hg) or <85 mm Hg, Diastolic BP >105 mm Hg, resting pulse rate: >120 bpm or <50 bpm, difference in systolic BP at Visit x (increase or decrease) compared with pretreatment >40 mm Hg and difference in pulse rate at Visit x (increase or decrease) compared with pretreatment >30 bpm. Baseline of double-blind treatment period was defined as the average of the measurements of the last 2 weeks at site prior to first intake of double-blind study medication.
Time Frame: Baseline period (Week -3 up to -1), treatment period (Baseline up to Week 56)
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Treatment Period: Ciclesonide 160 mcg | Treatment Period: Ciclesonide 320 mcg | Treatment Period: Ciclesonide 640 mcg
Number analyzed (Participants) | 119 | 122 | 126
participants | 0 | 0 | 0

13. Secondary Outcome: Number of Participants Reporting Clinically Significant Change From Baseline in Physical Examination Findings
Description: Physical examination consists of examinations of the following body systems: (1) eyes; (2) ears, nose, throat; (3) cardiovascular system; (4) respiratory system; (5) gastrointestinal system; (6) dermatologic system; (7) extremities; (8) musculoskeletal system; (9) nervous system; (10) lymph nodes; and (11) physical examinations other than body systems described in (1) to (10). Baseline of double-blind treatment period was defined as the average of the measurements of the last 2 weeks at site prior to first intake of double-blind study medication.
Time Frame: Baseline period (Week -3 up to -1), treatment period (Baseline up to Week 56)
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Treatment Period: Ciclesonide 160 mcg | Treatment Period: Ciclesonide 320 mcg | Treatment Period: Ciclesonide 640 mcg
Number analyzed (Participants) | 119 | 122 | 126
participants | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Markedly Abnormal Laboratory Values
Description: The number of participants with any markedly abnormal standard safety laboratory values collected throughout study. Baseline of double-blind treatment period was defined as the average of the measurements of the last 2 weeks at site prior to first intake of double-blind study medication.
Time Frame: Baseline period (Week -3 up to -1), treatment period (Baseline up to Week 56)
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Treatment Period: Ciclesonide 160 mcg | Treatment Period: Ciclesonide 320 mcg | Treatment Period: Ciclesonide 640 mcg
Number analyzed (Participants) | 119 | 122 | 126
participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 30 days for a serious adverse event after the last dose of double-blind study drug.
Description: Investigator documented any AEs and abnormal laboratory findings.Any event spontaneously reported was recorded,irrespective of the relation to study treatment.1 participant erroneously randomized into 160 mcg arm,actually received 640 mcg dose.For safety analysis,participants were analyzed based on the treatment they actually received.
Arm/Group | Baseline Period: Ciclesonide 160 mcg | Treatment Period: Ciclesonide 160 mcg | Treatment Period: Ciclesonide 320 mcg | Treatment Period: Ciclesonide 640 mcg
Serious Adverse Events (participants affected / at risk) | 1/520 | 6/119 | 9/122 | 0/126
Other Adverse Events (participants affected / at risk) | 64/520 | 65/119 | 65/122 | 70/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Baseline Period: Ciclesonide 160 mcg (N=520) | Treatment Period: Ciclesonide 160 mcg (N=119) | Treatment Period: Ciclesonide 320 mcg (N=122) | Treatment Period: Ciclesonide 640 mcg (N=126)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 2 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Invertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebellar ischaemia (Nervous system disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Baseline Period: Ciclesonide 160 mcg (N=520) | Treatment Period: Ciclesonide 160 mcg (N=119) | Treatment Period: Ciclesonide 320 mcg (N=122) | Treatment Period: Ciclesonide 640 mcg (N=126)
Bronchitis (Infections and infestations) | 1 | 18 | 16 | 16
Influenza (Infections and infestations) | 0 | 6 | 6 | 11
Nasopharyngitis (Infections and infestations) | 6 | 23 | 25 | 22
Pharyngitis (Infections and infestations) | 1 | 4 | 8 | 4
Rhinitis (Infections and infestations) | 6 | 2 | 8 | 4
Sinusitis (Infections and infestations) | 1 | 7 | 5 | 8
Upper respiratory tract infection (Infections and infestations) | 3 | 7 | 1 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 2 | 8
Headache (Nervous system disorders) | 43 | 22 | 23 | 16
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 7 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 7 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 8 | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.